CLINICAL TRIAL: NCT07100002
Title: Comparing the Efficacy of Earplugs and Eye Masks on Pain and Sleep Quality in Cardiovascular Intensive Care Unit Patients: A Three-Arm Randomized Controlled Trial
Brief Title: Comparing the Efficacy of Earplugs and Eye Masks on Pain and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Esra Ozkan, Assistant Prof., Giresun University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Giresun Üniversitesi
Record Dates: First submitted 2025-02-22; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Sleep Quality; Pain; Intensive Care Medicine; Cardiac Surgery
Keywords: Cardiac surgery, earplug, eye-mask, intensive care unit
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A Three-Arm Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator)
  Interventions: Device: Control Group
- Earplug Group (Experimental): Patients who met the inclusion criteria were fitted with standard earplug of the same brand by the researcher at night. The researcher applied the earplug from 01:00 AM to 05:00 AM. The reason for this is that the procedures performed on the patients within the clinical routine ended at 01:00 AM and the patients' uninterrupted sleep hours coincided with these hours.
  Interventions: Device: Earplug Group
- Eye mask Group (Experimental): Patients who met the inclusion criteria were fitted with standard eye masks of the same brand by the researcher at night. The researcher applied the eye mask from 01:00 AM to 05:00 AM. The reason for this is that the procedures performed on the patients within the clinical routine ended at 01:00 AM and the patients' uninterrupted sleep hours coincided with these hours.
  Interventions: Device: Eye mask Group

INTERVENTIONS:
Device: Control Group — Patients in this group did not receive any treatment to improve pain and sleep quality during the study period. Routine postoperative care was applied in the clinic.
  Arms: Control Group
Device: Earplug Group — Patients who met the inclusion criteria were fitted with standard earplug of the same brand by the researcher at night. The researcher applied the earplug from 01:00 AM to 05:00 AM. The reason for this is that the procedures performed on the patients within the clinical routine ended at 01:00 AM and the patients' uninterrupted sleep hours coincided with these hours.
  Arms: Earplug Group
Device: Eye mask Group — Patients who met the inclusion criteria were fitted with standard eye masks of the same brand by the researcher at night. The researcher applied the eye mask from 01:00 AM to 05:00 AM. The reason for this is that the procedures performed on the patients within the clinical routine ended at 01:00 AM and the patients' uninterrupted sleep hours coincided with these hours.
  Arms: Eye mask Group

SUMMARY:
Objective: To determine the superiority of earplugs and eye masks to each other and their efficacy in pain and sleep quality.

Methods: The study was a three-arm randomised controlled trial. After a baseline assessment, participants were randomly assigned in three groups. The random assignment was performed by using a computer program (Microsoft Excel 2016). Afterward, participants were categorized into three subgroups. Group 3 patients in this group did not receive any treatment to improve pain and sleep quality during the study period. Routine postoperative care was applied in the clinic (n = 25). Group 2 was applied the earplug (n = 25), whereas Group 1 was applied the eye mask (n = 24).

DETAILED DESCRIPTION:
Cardiovascular diseases are among the most common and leading causes of death worldwide. Surgical methods such as coronary artery bypass graft surgery (CABG) provide successful results in this process. (1) Patients who are faced with these disturbing life-threatening experiences try to cope with many problems until the discharge process. The most common of these problems in the postoperative period is pain. Incision in the sternal region, saphenous vein grafting and the presence of chest and mediastinal tubes are reported to cause pain in patients following cardiac surgery (2,3) Pain is an inevitable condition for many patients after surgery. Inappropriate pain control leads to activation of the sympathetic nervous system and increased hormonal responses to stress. It may also lead to decreased patient satisfaction, delayed mobilization and increased risk of deep vein thrombosis and pulmonary thromboembolism (2) Inadequate pain management causes sleep deprivation, exhaustion and disorientation as well as agitation, which are common in critically ill patients (4,5).It has been reported that adult patients receiving treatment in the intensive care unit (ICU)often complain of difficulty sleeping or frequent awakenings (6). Excessive noise, bright lights, frequent medical procedures, routine monitoring of vital signs, invasive devices, medications, pain, and anxiety in the ICU contribute to a reduction in sleep quality (7,8). Many systematic reviews provide evidence that earplugs and eye masks impact sleep quality and the incidence of delirium. However, the literature highlights a lack of high-quality studies to confirm these findings (6,14). It was also determined that there were studies to determine the effect of eyemask and earplugs on sleep and pain level (10,11,12), however, there are no studies examining the superiority of earplugs or eye masks over each other. For this reason, the research was carried out to determine the superiority of earplugs and eye masks to each other.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and older,
* Having undergone first and elective cardiac surgery, literate, and having no verbal communication skills.
* The participants who stayed in the ICU for 48 hours after surgery, had an ASA (American Society of Anesthesiologists) Score of I or II, and had no visual or audial problems were also included in the study.

Exclusion Criteria:

* Exclusion criteria for the study participants were refusing to use an eye mask or earplug, having early complications or re-surgery history, having reintubation after extubation, having any intra-aortic balloon pump or cardiac pacemaker, and taking inotropic drugs in the ICU.
* Patients refusing to use an eye mask or earplugs were also excluded from the study. Additionally, patients who had a history of chronic pain, alcohol or drug dependency, psychiatric disease, chronic sleep disorders, anxiolytic or sleeping medication use, and claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative sleep quality | 6 month
  Sleep quality was assessed using the Richard Campbell Sleep Questionnaire.
Postoperative pain severty | 6 month
  Pain was assessed using the Visual Analyses Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Giresun Universitesi, Giresun, Piraziz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33196559/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32006033/